CLINICAL TRIAL: NCT01267864
Title: IV Valproate for Acute Migraine. A Randomized Comparison Versus IV Metoclopramide and IV Ketorolac
Brief Title: Valproate Versus Ketorolac Versus Metoclopramide
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Principal Investigator, Benjamin W. Friedman, MD, Associate professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-01-009
Record Dates: First submitted 2010-12-15; First posted 2010-12-29 (Estimated); Results first posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Acute Migraine
Keywords: migraine; emergency; metoclopramide; ketorolac; valproate
MeSH Terms: conditions — Migraine Disorders; Emergencies | interventions — Metoclopramide; Ketorolac; Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Metoclopramide (Active Comparator): Metoclopramide 10mg IVSS
  Interventions: Drug: Metoclopramide
- Ketorolac (Active Comparator): Ketorolac 30mg IV
  Interventions: Drug: Ketorolac
- Valproate (Active Comparator): 1gm IV
  Interventions: Drug: Valproate

INTERVENTIONS:
Drug: Metoclopramide — 10mg IVSS
  Arms: Metoclopramide
Drug: Ketorolac — 30g IVSS
  Arms: Ketorolac
Drug: Valproate — 1gm IVSS
  Arms: Valproate

SUMMARY:
This randomized study is testing 3 different intravenous medications to see which one is best for acute migraine. The three medications are metoclopramide, valproate, and ketorolac.

DETAILED DESCRIPTION:
One million patients present to US emergency departments (ED) annually for treatment of acute migraine headache. A variety of parenteral medications are used to treat acute migraine, but none offer rapid and complete headache relief without side effects. Preliminary studies have suggested that intravenous valproate, an anti-epileptic medication with established efficacy as a migraine preventive, may be useful for the treatment of acute migraine. We propose a randomized, comparative efficacy trial in which intravenous valproate is compared to two standard parenteral therapies for acute migraine. There will not be a placebo control. Included subjects will be adults 64 years and younger who meet International Headache Society criteria for acute migraine, who do not have clinical evidence of secondary (organic) headache, and who do not have allergy or contra-indication to the investigational medications. The investigational medications are 1gm of valproate, 10mg of metoclopramide, and 30mg of ketorolac. Patients will be approached for participation and randomized at the time of presentation to the ED. Pain will be assessed on an 11 point (0 to 10) verbal pain scale, validated for use in acute pain trials. Medication will be infused as a slow intravenous drip. The primary outcome will be an improvement in headache intensity one hour after initiation of the intravenous drip. Secondary outcomes include assessments of pain, functional disability, adverse events, and satisfaction with the investigational medication one, two and 24 hours after initiation of the intravenous drip. The primary analysis will use a Student's t-test for independent samples and involve three pair-wise comparisons. Using an alpha of .017 (to account for the three pairwise comparisons), a standard beta, and a validated minimum clinically significant difference on the verbal pain scale, we calculated the need for 330 subjects. An interim analysis will be conducted to determine lack of efficacy of valproate.

ELIGIBILITY:
Inclusion Criteria:

* IHS migraine without aura
* IHS probable migraine (all migraine without arua criteria must be met except duration may be >72 hours or <4 hours)

Exclusion Criteria:

* Allergy or contra-indication to investigational medication

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 330 (Actual)
Dates: Start 2010-11; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Metoclopramide: Metoclopramide 10mg IVSS
  Metoclorpamide: 10mg IVSS
Period: Overall Study
Arm/Group | Metoclopramide | Ketorolac | Valproate
Started | 110 | 110 | 110
Completed | 110 | 110 | 110
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metoclopramide | Ketorolac | Valproate | Total
Number analyzed (Participants) | 110 | 110 | 110 | 330
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34 [26 to 44] | 34 [25 to 44] | 33 [25 to 41] | 33 [25 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 93 | 91 | 276
  Male | 18 | 17 | 19 | 54

OUTCOME MEASURES:

1. Primary Outcome: Headache Pain Level on a 0-10 Verbal Scale
Description: Verbal Numerical Rating scale for pain. Absolute change from baseline. This is a 0-10 scale on which 0= no pain and 10= the worst pain imaginable.
Time Frame: 60 minutes after receipt of medication
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Metoclopramide | Ketorolac | Valproate
Number analyzed (Participants) | 110 | 110 | 110
units on a scale | 4.7 [4.2 to 5.2] | 3.9 [3.3 to 4.5] | 2.8 [2.3 to 3.3]

2. Secondary Outcome: Participants Who Achieve Sustained Headache Freedom for 24 Hours
Description: Number of participants achieving a pain free state within two hours and maintaining the pain free state for 24 hours after receipt of medication
Time Frame: 2- 24 hours after receipt of medication
Population: Please note that 1 patient in the metoclopramide arm and 1 patient in the ketorolac arm were lost-to-follow-up and did not provide data for this outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Metoclopramide | Ketorolac | Valproate
Number analyzed (Participants) | 109 | 109 | 110
Participants | 12 | 17 | 4

3. Secondary Outcome: Satisfaction With Medication
Description: % who answer the following question affirmatively at 24 hours: Do you want to receive the same medication the next time you present to an ER with an acute migraine
Time Frame: 24 hours
Population: Study participants were telephoned 24 hours after medication administration. 3 patients in the metoclopramide arm, 4 in the ketorolac arm, and 3 in the valproate arm were lost to follow-up and did not provide these data. Additionally, 1 patient in the ketorolac arm did not provide an answer to this question
Measure: Count of Participants; unit: Participants
Arm/Group | Metoclopramide | Ketorolac | Valproate
Number analyzed (Participants) | 107 | 105 | 107
Participants | 65 | 42 | 28

4. Secondary Outcome: Adverse Event
Description: % who report any adverse event after administration of investigational medication
Time Frame: 24 hours
Population: Any adverse event reported at any assessment throughout the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | Metoclopramide | Ketorolac | Valproate
Number analyzed (Participants) | 109 | 110 | 110
Participants | 24 | 33 | 25

ADVERSE EVENTS:
Time Frame: Adverse events were assessed for two hours in the emergency department after medication administration and then by telephone 24 hours later.
Description: Please note: 3 patients in the metoclopramide arm, 5 in the ketorolac arm, and 3 in the valproate arm did not provide data about restlessness.
  Also, 1 patient in the metoclopramide arm did not provide any adverse event data.
  Please note: Patients who reported an adverse event but did not detail what their symptom was are counted as "other"
Arm/Group | Metoclopramide | Ketorolac | Valproate
Serious Adverse Events (participants affected / at risk) | 0/109 | 0/110 | 0/110
Other Adverse Events (participants affected / at risk) | 24/109 | 33/110 | 25/110
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metoclopramide (N=109) | Ketorolac (N=110) | Valproate (N=110)
Restless (Nervous system disorders) | 15 (15) | 10 (10) | 9 (9) — 24 hours after medication administration, we asked patients whether they had felt restless at any time after receiving the IV medication in the ED.
Drowsiness (Nervous system disorders) | 2 (2) | 2 (2) | 7 (7) — Too drowsy to function after receiving investigational medication
Dizzy (Nervous system disorders) | 8 (8) | 9 (9) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 1 | 4 | 2
Other (Investigations) | 15 (15) | 20 (20) | 17 (17) — Any other adverse event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes